CLINICAL TRIAL: NCT00647270
Title: A Multi-center, Randomized, Double-blind,Placebo-controlled Study Comparing 80 mg of Adalimumab With Placebo, and Demonstrating the Non-inferiority of Monthly 80 mg Adalimumab Dosing Compared With 40 mg Adalimumab Every Other Week Dosing
Brief Title: Study Comparing 80 mg of Adalimumab With Placebo, and Demonstrating the Non-inferiority of Monthly 80 mg Adalimumab Dosing Compared With 40 mg Adalimumab Every Other Week Dosing
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Beverly Paperiello, Director, Clinical Program Management, Abbott
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M10-261
Record Dates: First submitted 2008-03-27; First posted 2008-03-31 (Estimated); Results first posted 2010-05-10 (Estimated); Last update posted 2011-04-11 (Estimated); Status verified 2011-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo 12 weeks, 40mg adalimumab remaining 12 weeks
  Interventions: Drug: Placebo
- 40 mg (Active Comparator): 40 mg every other week
  Interventions: Drug: adalimumab
- 80 mg (Active Comparator): 80 mg monthly
  Interventions: Drug: adalimumab

INTERVENTIONS:
Drug: adalimumab — Pre-filled syringe. See arm for more detail
  Other Names: ABT-D2E7; Humira
  Arms: 40 mg
Drug: Placebo — Pre-filled syringe. See arm for more detail
  Arms: Placebo
Drug: adalimumab — Pre-filled syringe. See arm for more detail
  Other Names: ABT-D2E7; Humira
  Arms: 80 mg

SUMMARY:
To demonstrate the efficacy of 80 mg adalimumab monthly dosing compared with placebo and demonstrate the non-inferiority of monthly dosing of 80 mg adalimumab compared with dosing of 40 mg adalimumab every other week.

DETAILED DESCRIPTION:
The objective of this study is to demonstrate the efficacy of 80 mg adalimumab monthly dosing compared with placebo as measured by ACR20 response criteria following 12 weeks of therapy. The study is also designed to demonstrate the non-inferiority of monthly dosing of 80 mg adalimumab compared with dosing of 40 mg adalimumab eow as measured by ACR20 response criteria at Week 12.

ELIGIBILITY:
Inclusion Criteria:

* Subject > 18 years of age
* Subject has a diagnosis of RA as defined by the 1987-revised ACR-classification criteria and has a disease duration for a minimum of three months
* Subject must meet the following two criteria: a) At least 6 swollen joints out of 66 assessed, or b) At least 6 tender joints out of 68 assessed
* If a subject is on MTX, the doses must be stable for at least 4 weeks prior to Screening blood draw and follow standard recommendations for MTX treatment
* Subject is judged to be in generally good health as determined by the principal investigator

Exclusion Criteria:

* Subject has previous exposure to any systemic anti-TNF therapy (eg, infliximab, etanercept, certolizumab pegol or golimumab) including adalimumab
* Subject has a history of acute inflammatory joint disease of different origin other than RA
* Subject has been treated with any investigational biologic agents
* Subject considered by the investigator, for any reason, to be an unsuitable candidate for the study
* Female subject who is pregnant or breast-feeding or considering becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 2007-12; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Redden, MD, Study Director — Abbott
Locations (83):
- United States (47):
  - Huntsville, Alabama
  - Tuscaloosa, Alabama
  - Paradise Valley, Arizona
  - Hemet, California
  - Long Beach, California
  - Santa Monica, California
  - Torrance, California
  - Victorville, California
  - West Hills, California
  - Wheat Ridge, Colorado
  - Aventura, Florida
  - Orange Park, Florida
  - Palm Harbor, Florida
  - Sarasota, Florida
  - Tampa, Florida
  - Vero Beach, Florida
  - Atlanta, Georgia
  - Chicago, Illinois
  - Moline, Illinois
  - Springfield, Illinois
  - Wichita, Kansas
  - Lexington, Kentucky
  - Covington, Louisiana
  - Brighton, Michigan
  - Passaic, New Jersey
  - Smithtown, New York
  - The Bronx, New York
  - Ashville, North Carolina
  - Charlotte, North Carolina
  - Hickory, North Carolina
  - Monroe, North Carolina
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Bethlehem, Pennsylvania
  - Duncansville, Pennsylvania
  - Philadelphia, Pennsylvania
  - West Reading, Pennsylvania
  - Charleston, South Carolina
  - Greenville, South Carolina
  - Jackson, Tennessee
  - Nashville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Ogden, Utah
  - Olympia, Washington
  - Glendale, Wisconsin
- Australia (2):
  - Brisbane, Queensland
  - Cairns, Queensland
- Canada (16):
  - Winnipeg, Manitoba
  - Fredericton, New Brunswick
  - St. John's, Newfoundland and Labrador
  - Lunenburg, Nova Scotia
  - Burlington, Ontario
  - Hamilton, Ontario
  - Kitchener, Ontario
  - Newmarket, Ontario
  - Ottawa, Ontario
  - Saint Catherines, Ontario
  - Sarnia, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Québec, Quebec
  - Saint-Eustache, Quebec
  - Sainte-Foy, Quebec
- Germany (8):
  - Bad Nauheim
  - Berlin
  - Buch
  - Frankfurt
  - Freiburg im Breisgau
  - München
  - Würzburg
  - Zerbst
- Puerto Rico (2):
  - Caguas
  - Ponce
- United Kingdom (8):
  - Metropolitan Borough of Wirral, Cheshire
  - Liverpool, Merseyside
  - Oxford, Oxfordshire
  - Bath, Somerset
  - Cannock, Staffordshire
  - Newcastle upon Tyne, Tyne and Wear
  - Leeds, Yorkshire
  - Huddersfield, York

REFERENCES:
- [Derived] Burmester GR, Landewe R, Genovese MC, Friedman AW, Pfeifer ND, Varothai NA, Lacerda AP. Adalimumab long-term safety: infections, vaccination response and pregnancy outcomes in patients with rheumatoid arthritis. Ann Rheum Dis. 2017 Feb;76(2):414-417. doi: 10.1136/annrheumdis-2016-209322. Epub 2016 Jun 23. PMID 27338778

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 72 sites in the United States, Canada, Puerto Rico, Germany, the United Kingdom, and Australia. Subjects received over the course of 24 weeks either 80 mg adalimumab monthly, 40 mg adalimumab every other week (eow), or placebo (12 weeks) followed by 40 mg adalimumab eow (12 weeks).
Pre-assignment Details: A total of 432 subjects were enrolled, randomized, and received at least 1 dose of study drug. A total of 420 subjects were defined as the Full analysis set (FAS), which excluded the 12 subjects enrolled at a non-compliant site. A total of 48 subjects were switched from placebo to adalimumab 40 mg eow and participated in Period 2.
Groups:
- Placebo: Placebo 40 mg every other week (eow) for 12 weeks for Period 1; Adalimumab 40 mg eow for remaining 12 weeks for Period 2
- Adalimumab 40 mg Eow: Adalimumab 40 mg eow for Period 1 and Period 2
- Adalimumab 80 mg Monthly: Adalimumab 80 mg monthly for Period 1 and Period 2
Period: Period 1, Placebo-control (12 Weeks)
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Started | 56 (Placebo subjects in Period 1 received adalimumab 40 mg every other week in Period 2.) | 159 | 205
Completed | 48 | 146 | 182
Not Completed | 8 | 13 | 23
Not completed — Adverse Event | 2 | 7 | 7
Not completed — Lost to Follow-up | 0 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 7
Not completed — Other | 4 | 4 | 8
Period: Period 2, Placebo Switched to Adalimumab
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Started | 48 (Placebo subjects in Period 1 received adalimumab 40 mg eow in Period 2) | 146 | 182
Completed | 45 | 137 | 175
Not Completed | 3 | 9 | 7
Not completed — Adverse Event | 1 | 3 | 3
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Other | 2 | 6 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly | Total
Number analyzed (Participants) | 56 | 159 | 205 | 420
Age, Customized [Number; unit: participants]
  < 65 years | 43 | 113 | 148 | 304
  >= 65 years | 13 | 46 | 57 | 116
Age Continuous [Mean (Standard Deviation); unit: years] | 54.4 (12.46) | 57.2 (12.79) | 56.3 (12.43) | 56.4 (12.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 122 | 149 | 314
  Male | 13 | 37 | 56 | 106

OUTCOME MEASURES:

1. Primary Outcome: The Number of Responders According to the American College of Rheumatology (ACR) 20 Response Criteria at Week 12 Involving the Comparison of Adalimumab 80 mg Monthly Dose Versus Placebo and Adalimumab 40 mg Every Other Week (Eow)
Description: Comparison of adalimumab 80 mg monthly dose versus placebo and adalimumab 40 mg eow in the number of responders with ACR criteria improvement consisting of 20%, (ACR20) reduction in tender or swollen joint counts (TJC or SJC, respectively) and 20% improvement in 3 of the following 5 criteria: [1] physician's global assessment of disease activity (PGA), [2] subject's assessment of disease activity, [3] subject's assessment of pain, [4] subject's assessment of physical disability via a health assessment questionnaire disability index(HAQ-DI), and [5] C-reactive protein (CRP) at each visit
Time Frame: Week 12
Population: Full Analysis Set (FAS) - a subset of the intent to treat population used in all efficacy analyses excluding subjects from an Abbott identified Investigator who was non-compliant with the protocol requirements. The FAS of subjects who received at least 1 dose of study drug during Period 2 of the study was used for Period 2 efficacy analyses.
Measure: Number; unit: participants
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Number analyzed (Participants) | 56 | 159 | 205
participants
  Responders | 19 | 80 | 97
  Nonresponders | 37 | 79 | 108
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80 mg Monthly; Adalimumab 80 mg monthly versus placebo: The null hypothesis associated with this comparison stated that adalimumab 80 mg monthly would be inferior to placebo with respect to ACR20 response percentage; the alternative hypothesis was that adalimumab 80 mg monthly would be superior to placebo with respect to ACR20 response; Test type: Superiority or Other; p = 0.074, Chi-squared; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-13.3 to 7.4] — Treatment difference between adalimumab 80 mg monthly and placebo divided by the difference between adalimumab 40 mg eow and placebo
Statistical Analysis 2: Comparison: Adalimumab 40 mg Eow vs Adalimumab 80 mg Monthly; The non-inferiority of adalimumab 80 mg monthly to adalimumab 40 mg every other week (eow) was to be claimed if at least 50% of the treatment effect of adalimumab 40 mg eow over placebo was to be achieved by adalimumab 80 mg monthly over placebo; Test type: Non-Inferiority or Equivalence — A sensitivity analysis was proposed for the non-inferiority comparison. If the lower confidence limit of θ80 - θ40 was greater than -0.1, then the non-inferiority of adalimumab 80 mg monthly to adalimumab 40 mg eow would be claimed; p = 0.74, Chi-squared — Non - inferiority of adalimumab 80 mg monthly compared with 40 mg eow could not be tested because the null hypothesis of the first comparison was not rejected

2. Secondary Outcome: Within Group Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Observed)
Description: The HAQ-DI is a self-reported subject measure of physical function calculated as the mean of 8 category scores: Dressing and Grooming, Rising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Each category score is calculated as the maximum of the scores for the questions within the category. The HAQ-DI is expressed on a scale of 0 (without any difficulty) to 3 (unable to do) representing an average score across the category. Scores for at least 6 categories are needed to compute the HAQ score. Changes to lower scores indicate improvement in physical function.
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS)-a subset of the intent to treat population used in all efficacy analyses excluding subjects from an Abbott identified Investigator who was non-compliant with protocol requirements. The FAS of subjects who received at least 1 dose of study drug during Period 2 of the study was used for Period 2 efficacy analyses (observed).
Measure: Mean (Standard Deviation); unit: units on a score
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Number analyzed (Participants) | 56 | 159 | 205
units on a score | -0.11 (0.488) | -0.41 (0.508) | -0.39 (0.536)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80 mg Monthly; Using a fixed-sequence multiple-testing approach at an alpha level of 0.05 to test the secondary endpoints, the testing of the null-hypothesis began with the first endpoint and stopped as soon as failure to reject a hypothesis occurred (i.e., P value > 0.05). Using this procedure, testing stopped after secondary endpoint number 1, change from Baseline in HAQ at Week 12; Test type: Superiority or Other; p = 0.002, ANCOVA

3. Secondary Outcome: Within Group Mean Change From Baseline in the Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Last Observation Carried Forward [LOCF])
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: Full Analysis Set (FAS)-a subset of the intent to treat population used in all efficacy analyses excluding subjects from an Abbott identified Investigator who was non-compliant with protocol requirements. The FAS of subjects who received at least 1 dose of study drug during Period 2 of the study was used for Period 2 efficacy analyses (LOCF).
Measure: Mean (Standard Deviation); unit: units on a score
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Number analyzed (Participants) | 56 | 159 | 205
units on a score | -0.12 (0.484) | -0.40 (0.507) | -0.37 (0.537)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80 mg Monthly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA
Statistical Analysis 2: Comparison: Placebo vs Adalimumab 40 mg Eow; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA

4. Secondary Outcome: Between Group Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Observed)
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a score
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Number analyzed (Participants) | 56 | 159 | 205
units on a score | 0 (0) | -0.26 (0.081) | -0.24 (0.079)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 40 mg Eow vs Adalimumab 80 mg Monthly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.002, ANCOVA — The ANCOVA Model was adjusted for the Baseline Measure

5. Secondary Outcome: Between Group Mean Change From Baseline in Health Assessment Questionnaire Disability Index (HAQ-DI) at Week 12 (Last Observation Carried Forward [LOCF])
Description: as for outcome 2
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a score
Arm/Group | Placebo | Adalimumab 40 mg Eow | Adalimumab 80 mg Monthly
Number analyzed (Participants) | 56 | 159 | 205
units on a score | 0 (0) | -0.24 (0.077) | -0.21 (0.075)
Statistical Analysis 1: Comparison: Placebo vs Adalimumab 80 mg Monthly; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.005, ANCOVA — The ANCOVA Model was adjusted for Baseline Measure; The ANCOVA Model was adjusted for Baseline Measure

ADVERSE EVENTS:
Time Frame: 24 Weeks
Groups:
- Placebo Every Other Week (Eow)-Period 1: Placebo eow for 12 weeks for Period 1 Adalimumab 40 mg eow for remaining 12 weeks for Period 2
- Adalimumab 40 mg Eow -Period 1; Adalimumab 40 mg Eow-Period 2: Adalimumab 40 mg eow for Period 1 and Period 2
- Adalimumab 80 mg Monthly-Period 1; Adalimumab 80 mg Monthly - Period 2: Adalimumab 80 mg monthly for Period 1 and Period 2
- Placebo/Adalimumab 40 mg Eow-Period 2: Placebo 40 mg eow for Period 1 (weeks 1-12) Subjects switched to Adalimumab 40 mg eow for remaining 12 weeks for Period 2
Arm/Group | Placebo Every Other Week (Eow)-Period 1 | Adalimumab 40 mg Eow -Period 1 | Adalimumab 80 mg Monthly-Period 1 | Placebo/Adalimumab 40 mg Eow-Period 2 | Adalimumab 40 mg Eow-Period 2 | Adalimumab 80 mg Monthly - Period 2
Serious Adverse Events (participants affected / at risk) | 5/57 | 8/164 | 4/211 | 1/49 | 5/151 | 12/188
Other Adverse Events (participants affected / at risk) | 13/57 | 29/164 | 38/211 | 6/49 | 14/151 | 11/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Every Other Week (Eow)-Period 1 (N=57) | Adalimumab 40 mg Eow -Period 1 (N=164) | Adalimumab 80 mg Monthly-Period 1 (N=211) | Placebo/Adalimumab 40 mg Eow-Period 2 (N=49) | Adalimumab 40 mg Eow-Period 2 (N=151) | Adalimumab 80 mg Monthly - Period 2 (N=188)
Abdominal adhesions (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Small intestinal stenosis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 2 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Meningitis meningococcal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 4 | 0 | 0 | 1 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Patella fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Pubic rami fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Myocardial infaection (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Death (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Meningitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Splenic haematoma (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalamia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Every Other Week (Eow)-Period 1 (N=57) | Adalimumab 40 mg Eow -Period 1 (N=164) | Adalimumab 80 mg Monthly-Period 1 (N=211) | Placebo/Adalimumab 40 mg Eow-Period 2 (N=49) | Adalimumab 40 mg Eow-Period 2 (N=151) | Adalimumab 80 mg Monthly - Period 2 (N=188)
diarrhoea (Gastrointestinal disorders) | 4 | 2 | 4 | 0 | 0 | 0
nausea (Gastrointestinal disorders) | 3 | 9 | 13 | 0 | 0 | 0
nasopharyngitis (Infections and infestations) | 3 | 8 | 2 | 3 | 10 | 5
upper respiratory tract infection (Infections and infestations) | 4 | 5 | 11 | 3 | 4 | 6
dizziness (Nervous system disorders) | 3 | 4 | 5 | 0 | 0 | 0
headache (Nervous system disorders) | 3 | 8 | 10 | 0 | 0 | 0
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Abbott identified Investigator non-compliance with the protocol requirements at one site and made the decision to exclude the data from this site from all efficacy analyses. Sample size was too small to demonstrate superiority and non-inferiority.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.